CLINICAL TRIAL: NCT02970006
Title: Investigating Mechanisms Underlying Spinal Cord Stimulation Efficacy Using Virtual Reality and Full Body Illusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Swiss Federal Institute of Technology (Other)
Responsible Party: Principal Investigator, Vibhor Krishna, Assistant Clinical Professor, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016H0202
Record Dates: First submitted 2016-11-16; First posted 2016-11-21 (Estimated); Results first posted 2021-09-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-08

CONDITIONS: Neuropathy;Peripheral
Keywords: spinal cord stimulation; virtual reality; full body illusion
MeSH Terms: conditions — Neuritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- neurovisual stimulation (Experimental): Participants in this study will be adults who have already undergone implantation of SCS for the treatment of their pain conditions. The study involves no further treatment or intervention. Subjects will be approached for participation in this study during their routine postoperative clinical visit to the Center for Neuromodulation at the Ohio State University (OSU).All eligible patients will undergo a one-day visit for the virtual reality and full body illusion intervention. This research will also investigate leg embodiment and leg analgesic effects during SCS integrated with different patterns of virtual leg illumination.
  Interventions: Device: neurovisual stimulation

INTERVENTIONS:
Device: neurovisual stimulation — a new system of multisensory stimulation based on virtual and enhanced reality (i.e., neuro-visual stimulation)

SUMMARY:
The study hypothesis is that spinal cord stimulation (SCS) combined with virtual leg illumination (provided through a wearable headset (OculusRift, OculusVR, Irvine, CA) and a custom-designed virtual reality leg scenario) will lead to controlled analgesia induction, boosting analgesic effects obtained with standard SCS treatments and will further be associated with changes in the perception of the affected body part.

DETAILED DESCRIPTION:
Epidural spinal cord stimulation (SCS) is an approved treatment for truncal and extremity neuropathic pain. The mechanisms underlying the efficacy of SCS are unknown. Recent advances in cognitive neuroprosthetics using virtual reality allow for modulation of body perception and bodily experience, which has also been shown to modulate pain perception. The present research proposal plans to merge expertise in cognitive neuroprosthetics with neuromodulation techniques in order to test the analgesic properties of the combination of epidural spinal cord stimulation with a new system of multisensory stimulation based on virtual and enhanced reality (i.e., neuro-visual stimulation). The investigators propose to study this hypothesis prospectively in 25 patients with implanted SCS systems for the treatment of chronic neuropathic pain. Primary outcomes will be pain reduction (based on subjective, functional and physiological measures) and changes in body perception (based on subjective and objective measures). The present study will generate a proof-of-concept for the application of neuro-visual stimulation for the treatment of chronic pain and will form the basis for future NIH funding application.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-and older at the time of enrollment
2. Patients carrying a diagnosis of CPRS type 125 or chronic refractory neuropathic leg pain following FBS4
3. Patients who have implanted epidural SCS
4. The SCS implantation for at least three months prior to enrollment
5. Patients with efficacious SCS as defined by ≥ 50% pain improvement after switching SCS from an OFF state to an ON state ('optimal' stimulation efficacy)
6. Patients willing and able to provide informed consent

Exclusion Criteria:

1. Patients who are unable to effectively or efficiently communicate for example patients suffering from speech deficits (dysarthria, aphasia) or are non-English speaking.
2. Patients with history of prior cranial surgery, significant brain lesions for example intracranial tumors, strokes etc.
3. Non efficacious response to SCS <50% pain improvement with optimal stimulation parameters
4. Evidence of untreated psychiatric disorders or drugs/alcohol abuse.
5. History of seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2019-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vibhor R Krishna, MBBS, Principal Investigator — Ohio State University
Locations (1):
- The Ohio Sate University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Solca M, Krishna V, Young N, Deogaonkar M, Herbelin B, Orepic P, Mange R, Rognini G, Serino A, Rezai A, Blanke O. Enhancing analgesic spinal cord stimulation for chronic pain with personalized immersive virtual reality. Pain. 2021 Jun 1;162(6):1641-1649. doi: 10.1097/j.pain.0000000000002160. PMID 33259460

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Neurovisual Stimulation
Started | 15
Completed | 14
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Neurovisual Stimulation
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (9.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Average Pain Reduction Post Intervention
Description: 10 point Visual Analog pain rating Scale. Subjective pain perception will be measured by pain ratings on a 10cm visual continuous analog scale (VAS). Patients rate their pain, ranging from "no pain" (bottom part of the scale) to "the worst imaginable pain" (upper part of the scale) (Huskisson 1974). The pain reduction will be an average total of the pain scores taken at hours 1, 2, 3, 4, and 5.
Time Frame: At each hour from 1-5 hours post intervention
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Neurovisual Stimulation
Number analyzed (Participants) | 14
score on a scale | 2.72 (0.6)

2. Secondary Outcome: Pain Reduction Base on Patient Perception
Description: Validated questionnaires developed by the collaborators (Swiss Federal Institute of Technology) will be used in order to investigate induced changes in leg perception and ownership. In particular, we will assess: 1) feeling of ownership towards the leg shown in the virtual reality set-up (leg ownership); 2) tactile sensations felt on the virtual legs, depending on the different conditions of SCS and visual stimulation. Patients will be asked to indicate how much they agreed with each item using a 7-point colored vertical Likert scale ranging from 0 (complete disagreement, the bottom extreme, red point) to +6 (complete agreement, the top extreme, green point).
Time Frame: per minute in each virtual reality condition for 10 minutes in each reality condition.
Population: Patients will rate their pain reduction on a scale of 0-6, each minute in each of the three virtual reality conditions. The pain score change reported is an average of all time points in all virtual reality settings. A change in pain rating was calculated between different SCS and VR conditions. Percentage pain reduction was then calculated to test whether SCS combined with VR reduced pain more significantly than VR alone. The calculation done was a mean score of all pain ratings at all points.
Measure: Mean (Standard Error); unit: average score on scale of pain reduction
Arm/Group | Neurovisual Stimulation
Number analyzed (Participants) | 15
average score on scale of pain reduction | 0.7 (0.25)

ADVERSE EVENTS:
Time Frame: The experiment included 2 sessions occurring at 24 hours interval, the first session was used for clinical assessment and the personalization of the visual illumination administered in the virtual environment, while the experimental protocol was performed the second day. The duration of each session was between 90-120 minutes. Adverse events were monitored over that time.
Arm/Group | Neurovisual Stimulation
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2017-07-08): https://cdn.clinicaltrials.gov/large-docs/06/NCT02970006/Prot_000.pdf